CLINICAL TRIAL: NCT03047174
Title: Radiotherapy Related Skin Toxicity: Mepitel® Film vs. Standard Care in Patients With Locally Advanced Head-and-Neck Cancer
Brief Title: Radiotherapy Related Skin Toxicity: Mepitel® vs. Standard Care in Patients With Locally Advanced Head-and-Neck Cancer
Acronym: RAREST-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Prof. Dirk Rades, MD, Professor Dr. med., University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RAREST-01
Record Dates: First submitted 2017-01-26; First posted 2017-02-08 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and Neck Neoplasms, Radio(chemo)therapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Treatment with Mepitel® Film (Experimental): Arm A:
  Mepitel® Film is a gentle, sterile, transparent, breathable film dressing consisting of polyurethane film coated with a special contact layer. The film dressing is supported with a paper frame for ease of application. Mepitel® Film is an ultra thin, transparent, breathable soft silicone film dressing.
  Interventions: Other: Mepitel® Film
- Arm B: Treatment with Standard Care (Active Comparator): Cream: Fatty cream with 2-5% urea is applied to the irradiated skin 3-4 times daily.
  Mometasone furoate cream: In addition to the fatty cream with 2-5% urea, mometasone furoate cream (solution 0.1%) is applied to the irradiated skin once daily.
  Mometasone furoate cream is used in the treatment of inflammatory skin disorders. In terms of steroid strength, it is more potent than hydrocortisone, and less potent than dexamethasone. It reduces inflammation by causing several effects such as reversing the activation of inflammatory proteins, activating the secretion of anti-inflammatory proteins, stabilizing cell membranes, and decreasing the influx of inflammatory cells. The exact anti-inflammatory mechanism of action is unknown.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Mepitel® Film — Mepitel® Film is a gentle, sterile, transparent, breathable film dressing consisting of polyurethane film coated with a special contact layer. The film dressing is supported with a paper frame for ease of application. Mepitel® Film is an ultra thin, transparent, breathable soft silicone film dressing.
  Arms: Arm A: Treatment with Mepitel® Film
Other: Standard Care — Cream: Fatty cream with 2-5% urea is applied to the irradiated skin 3-4 times daily.
  Mometasone furoate cream: In addition to the fatty cream with 2-5% urea, mometasone furoate cream (solution 0.1%) is applied to the irradiated skin once daily.
  Arms: Arm B: Treatment with Standard Care

SUMMARY:
The aim for the present study named RAREST (RAdiotherapy RElated Skin Toxicity) is to compare the new dressing with the standard skin care. 168 patients receiving radiotherapy alone or radiochemotherapy for locally advanced head-and-neck cancer will be included. The primary aim is to investigate the rate of patients experiencing severe, stressful radiation dermatitis. The skin status will daily be inspected and assessed by specially trained doctors and nursing staff.

It is expected that the new self-adhesive dressing is superior to standard care with respect to prevention of grade ≥2 radiation dermatitis in patients receiving radiotherapy or radio(chemo)therapy for a head-and-neck tumor. Thus, the dressing would be well qualified to become a new standard procedure at the skin care of patients with a head-neck tumor.

DETAILED DESCRIPTION:
The primary goal of this randomized trial is to demonstrate that Mepitel® Film is superior to Standard Care with respect to prevent grade ≥2 radiation dermatitis (RD) in patients receiving radio(chemo)therapy up to 50 Gy for locally advanced squamous cell carcinoma of the head-and-neck (SCCHN).

The primary aim of this randomized multinational multicenter trial is to investigate the rate of patients experiencing grade ≥2 RD (CTCAE v4.03) until 50 Gy of radiotherapy (RT).

Evaluation until 50 Gy of RT is the primary endpoint, since up to 50 Gy, the irradiated volume includes the primary tumor and the bilateral cervical and supraclavicular lymph nodes, and, therefore, is almost identical in all patients. After 50 Gy, the irradiated volume is much more individual, depending on location and size of the primary tumor, involvement of lymph nodes, and the treatment approach (definitive vs. adjuvant).

This is a randomized, active-controlled, parallel-group trial, comparing the following treatments of radiation related skin toxicity in patients with head-and-neck cancer:

Mepitel® Film (Arm A) vs. Standard Care (Arm B). About 4 contributing centers are planned to include an average of 21 patients/year. The recruitment duration of 168 patients = 24 months. The follow-up period will be 3 weeks. The total running time = 25 months.

Stratification by prognostic factors:

1. Tumor site: oropharynx/oral cavity vs. hypopharynx/larynx
2. Treatment approach: radiochemotherapy vs. RT alone
3. Participating site In case of very small groups due to uneven distribution of stratification groups, strata might be connected for Analysis (before data base lock and final analysis of the data).

This trial is for patients receiving definitive or adjuvant radio(chemo)therapy for locally advanced (SCCHN).

Radiotherapy RT is administered using conventional fractionation (5 x 2.0 Gy per week). In all patients, the initial target volume includes the region of the primary tumor plus bilateral cervical and supraclavicular lymph nodes up to 50 Gy.

Patients treated with adjuvant RT following complete resection of the primary tumor and the involved lymph nodes (R0-resection) receive a radiation boost of 10 Gy (5 x 2.0 Gy per week) to the regions of the primary tumor and the involved lymph nodes.

In case of a microscopically incomplete resection (R1-resection), the boost dose to the primary tumor region is 16 Gy.

In case of extra-capsular spread (ECS) of lymph nodes, the lymph nodes showing ECS receive an additional boost of 6 Gy (i.e. a cumulative boost dose of 16 Gy).

Patients receiving definitive RT, receive a boost of 10 Gy (5 x 2.0 Gy/week) to the primary tumor, the involved lymph nodes, and the lymph node levels adjacent to the involved lymph nodes. An additional boost of another 10 Gy (5 x 2.0 Gy/week) is administered to the primary tumor and the involved lymph nodes.

Treatment should be performed as either intensity-modulated RT (IMRT) or volumetric modulated arc therapy (VMAT) RT.

The rate of patients experiencing grade ≥2 RD (CTCAE v4.03) until the 5. week of therapy (50 Gy) is in focus of this clinical study. Additionally another 2 weeks of RT (up to 70 Gy) might be performed. This further treatment will be conducted in accordance with common treatment guidelines. The treatment of the patients > 50 Gy will not be analyzed within this study. The occurrence of adverse events (AEs) and serious adverse events (SAEs) will be documented for the duration of RT. The final dose of RT will be documented in the Case Report Form (CRF).

Concomitant Chemotherapy In patients who receive definitive RT, concomitant chemotherapy with cisplatin or carboplatin is administered. The cumulative cisplatin or carboplatin dose at the end of the 5. week of RT (50 Gy) should be 200 mg/m2. This cumulative dose may either be achieved with 20 mg/m2 given with RT fractions 1-5 and 21-25, 25 mg/m2 given with RT fractions 1-4 and 21-24, or weekly doses of 40 mg/m2.

Cisplatin or carboplatin will be administered after saline hydration as intravenous bolus infusion. The saline hyper-hydration will be given according to the investigational centre's routine. All patients treated with cisplatin or carboplatin in addition to RT must receive adequate anti-emetic therapy prior to the administration of cisplatin or carboplatin. It is recommended that a 5-Hydroxytryptamine type 3 (5HT3) antagonist (e.g. granisetron) and dexamethasone 8 mg i.v. are administered prior to each cycle of treatment.

Quality assurance plan:

Monitoring: The Center for Clinical Studies (ZKS) Lübeck will conduct clinical on-site monitoring at the German sites according to common guidelines and regulations.

According to SOPs, all trial specific monitoring activities will be defined before starting the trial and documented in writing (monitoring manual).

Patient registration and randomization The patients will be assigned two code numbers: the number of the contributing center plus a patient identification (ID) number, continuously ascending, starting with 001.

After registration, patients will be randomized in a 1:1 ratio to receive either Mepitel® Film (Arm A) or Standard Care (Arm B) for treatment of radiation related skin toxicity.

A stratified randomization will be performed in blocks. The stratification will be conducted for about 4 centers, 2 treatment approaches, 2 tumor sites.

The randomization will be performed centrally at the ZKS via fax. The proceeding is based on standard operating procedures (SOPs) of the ZKS. .

Sample size calculation The primary goal of this randomized trial is to demonstrate that Mepitel® Film is superior to Standard Care with respect to prevent grade ≥2 RD in patients receiving radio(chemo)therapy up to 50 Gy for locally advanced SCCHN.

The null hypothesis of equal rates of grade ≥2 skin toxicity is tested against the two-sided alternative hypothesis of different rates. Based on this hypothesis system, the sample size required for this trial is calculated taking into account the following assumptions:

* A Chi-square Test will be applied
* The two-sided significance level is set to 5%
* In patients treated with radio(chemo)therapy for locally advanced SCCHN, previous studies have suggested rates of grade ≥2 skin toxicity of 86-92% if standard skin care was administered.
* Based on these data, a rate of grade ≥2 skin toxicity of 85% can be assumed in the reference group ("worst-case"), i.e. in patients receiving standard care for skin toxicity.
* Administration of Mepitel® Film will be considered to be clinically relevant, if the rate of grade ≥2 skin toxicity can be reduced to 65%.
* The power to yield statistical significance if the the difference in rates is in fact 20 percentage points is set to 80%.

Based on these assumptions, 80 patients are required per study arm within the Full Analysis Set (FAS). Taking into account that 5% of patients will not qualify for FAS, a total of 168 patients should be randomized.

Statistical analysis General Considerations All data recorded in the CRFs describing the study population, toxicity and quality of life (QoL) will be analyzed descriptively. Categorical data will be presented in contingency tables with frequencies and percentages. Continuous data will be summarized with at least: frequency (n), median, quartiles, mean, SD, min and max. Number of patients with protocol deviations and listings describing the deviations will be provided.

In general, chi-square tests will be used to compare percentages in a two-by-two contingency table, replaced by Fisher´s exact test if the expected frequency in at least one cell of the associated table is less than 5. Stratified two-by-two contingency tables will be analyzed using Cochran-Mantel-Haenszel tests. Logistic regression models serve as multivariable methods for binary endpoint data. Comparison of ordinal variables between treatment arms will be performed using the asymptotic Wilcoxon-Mann-Whitney test, replaced by its exact version in case of ordinal categories with small number of categories and/or sparse data within categories. Any shift in location of quantitative variables between study groups will be performed with Wilcoxon-Mann-Whitney tests as well.

Time-to-event data will be analyzed by Kaplan-Meier methods, when merely non-informative censoring occurs. For statistical comparison, the logrank-test will be provided supplemented by multivariate Cox proportional hazards models.

The data analysis will be performed according to the statistical analysis plan (SAP), finalised prior to database lock and prior to statistical analysis.

Primary Endpoint The rates of patients experiencing grade ≥2 RD in patients receiving radio(chemo)therapy up to 50 Gy will be statistically compared using the Cochran-Mantel-Haenszel Chi-square test on a two-sided significance level of 5%. This test is the natural non-parametric extension of the Chi-square test for testing the treatment effect, while adjusting for the effects of the stratification variables used for randomization. For further assessment of the robustness of the results, a logistic regression model for grade ≥2 RD will be applied including the parameters used for stratification. In addition, a model including also additional patient characteristics will be fitted.

The confirmatory evaluation will be performed within the FAS, the Per Protocol Set serves for further sensitivity analyses.

Secondary endpoints Time to grade 2 RD until 50 Gy of RT is defined as the time from start of RT to at least grade 2 RD. Patients without grade 2 RD will be censored after the date of receiving a total dose of 50 Gy.

The distribution of the time to grade 2 RD until administration of 50 Gy will be described using Kaplan-Meier methods. These analyses will be stratified by treatment arm and prognostic risk groups used for randomization. Estimates of median time to grade 2 RD and estimates of rates for specific time points will be extracted from the Kaplan-Meier analyses together with the associated 95% confidence limits. The treatment differences will be tested using a stratified log-rank test, stratified by stratification factors. Furthermore, Cox proportional hazards models will be applied to yield adjusted estimates of the associated hazard ratios.

All other AEs as reported according to CTCAE v4.03 will also be subjected to statistical analysis. AE tables will present the total number of patients reporting at least one specific event and the maximum CTCAE grade. Patients reporting more than one episode of the same event will be counted only once by the worst CTCAE grade per patient. Special tables will be given for CTCAE Grade III/IV/V AEs. Analysis will be restricted to treatment related AEs and treatment related CTCAE Grade III/IV/V events.

QoL will be evaluated using the validated EORTC quality of life questionnaire (QLQ)-C30 and EORTC QLQ-H&N35 questionnaires. Data will be scored according to the algorithm described in the respective scoring manuals. For all QoL domains and items, descriptive analyses will be presented stratified by visit and treatment arm.

For descriptive statistical analysis, summary tables will be provided showing measures of location and dispersion (min, quartiles, median, max, mean, SD) stratified by visit, treatment arm. Individual score items will be subjected to statistical analysis. Absolute changes of QoL-scores from baseline will be tabulated stratified by treatment group and visit. For graphical illustrations, Box-Whisker diagrams will be presented across visits for each treatment group. Nonparametric (exact) Wilcoxon-Mann-Whitney tests will be applied for exploratory comparison purposes. Additional details of the QoL analysis will be described in the SAP.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven locally advanced squamous cell carcinoma of the head-and-neck (SCCHN)
* Conventionally fractionated (5x2 Gy per week) definitive or adjuvant radio(chemo)therapy
* Age ≥18 years
* Written informed consent
* Capacity of the patient to contract

Exclusion Criteria:

* N3 stage (lymph nodes >6 cm)
* Distant metastases (M1)
* Pregnancy, Lactation
* Treatment with epidermal growth factor receptor (EGFR)-antibodies (either given or planned)
* Expected non-compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Rades, Prof. Dr., Principal Investigator — Dep. of Radiation Oncology, Univ. of Lübeck, Univ. Med. Center S-H, Germany
Locations (2):
- Germany (2):
  - Department of Radiotherapy (Radiooncology), Christian-Albrechts-Universität zu Kiel and University Medical Center Schleswig-Holstein Campus Kiel, Kiel, Schleswig-Holstein
  - Department of Radiation Oncology, University of Lübeck and University Medical Center Schleswig-Holstein, Lübeck

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rades D, Narvaez CA, Splettstosser L, Domer C, Setter C, Idel C, Ribbat-Idel J, Perner S, Bartscht T, Olbrich D, Schild SE, Carl J. A randomized trial (RAREST-01) comparing Mepitel(R) Film and standard care for prevention of radiation dermatitis in patients irradiated for locally advanced squamous cell carcinoma of the head-and-neck (SCCHN). Radiother Oncol. 2019 Oct;139:79-82. doi: 10.1016/j.radonc.2019.07.023. Epub 2019 Aug 17. PMID 31431372
- [Derived] Narvaez C, Doemer C, Idel C, Setter C, Olbrich D, Ujmajuridze Z, Carl JH, Rades D. Radiotherapy related skin toxicity (RAREST-01): Mepitel(R) film versus standard care in patients with locally advanced head-and-neck cancer. BMC Cancer. 2018 Feb 17;18(1):197. doi: 10.1186/s12885-018-4119-x. PMID 29454311

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Treatment With Mepitel® Film: Mepitel® Film is a gentle, sterile, transparent, breathable film dressing consisting of polyurethane film coated with a special contact layer. The film dressing is supported with a paper frame for ease of application. Mepitel® Film is an ultra thin, transparent, breathable soft silicone film dressing.
  Mepitel® Film: Mepitel® Film is a gentle, sterile, transparent, breathable film dressing consisting of polyurethane film coated with a special contact layer. The film dressing is supported with a paper frame for ease of application. Mepitel® Film is an ultra thin, transparent, breathable soft silicone film dressing.
- Arm B: Treatment With Standard Care: Cream: Fatty cream with 2-5% urea is applied to the irradiated skin 3-4 times daily. Mometasone furoate cream: In addition to the fatty cream with 2-5% urea, mometasone furoate cream (solution 0.1%) is applied to the irradiated skin once daily.
Period: Overall Study
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care
Started | 28 | 29
Completed | 9 | 27
Not Completed | 19 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Customized [Count of Participants; unit: Participants]
  Age: <=62 years | 15 | 14 | 29
  Age: >=63 years | 13 | 15 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 22 | 24 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 28 | 29 | 57
Region of Enrollment [Number; unit: participants]
  Germany | 28 | 29 | 57
Tumor site [Count of Participants; unit: Participants]
  Oropharynx | 13 | 11 | 24
  Oral cavity | 4 | 6 | 10
  Hypopharynx | 5 | 7 | 12
  Larynx | 6 | 5 | 11
Tumor stage (American Joint Committee on Cancer) [Count of Participants; unit: Participants] — For assessment of the tumor stage, the folllwoing classification was used (American Joint Committee on Cancer):
  Stage I: T1NoMo Stage II: T2NoM0 Stage III: T1-3N1M0, T3N0M0 Stage IV: T1-3N2M0, T4aN0-2M0 (IVa); T1-4N3M0, T4bN0-3M0 (IVb); T1-4N0-3M1 (IVc)
  A higher stage is associated with a worse prognosis.
  Participants
    Stage II | 3 | 2 | 5
    Stage III | 7 | 7 | 14
    Stage IV | 18 | 20 | 38
Histologic grading [Count of Participants; unit: Participants] — For the histologic grading, the following classification was used:
  GX Grade cannot be assessed G1 Well differentiated (Low grade) G2 Moderately differentiated (Intermediate grade) G3 Poorly differentiated (High grade) G4 Undifferentiated (High grade)
  A higher grade is generally associated with a worse prognosis.
  Participants
    G 1-2 | 17 | 16 | 33
    G 3 | 9 | 12 | 21
    Gx | 2 | 1 | 3
Human papilloma virus (HPV) status [Count of Participants; unit: Participants]
  Negative | 18 | 16 | 34
  Positive | 8 | 10 | 18
  Unknown | 2 | 3 | 5
Surgery prior to radiotherapy [Count of Participants; unit: Participants]
  No | 13 | 15 | 28
  Yes | 15 | 14 | 29
Eastern Cooperative Oncology Group performance score [Count of Participants; unit: Participants] — Performance status was rated with the Eastern Cooperative Oncology Group (ECOG), ranging from 0 to 5 (lower grade=better performance status).
  0: Fully active without restrictions.
  1. Restricted in physically strenuous activity; ambulatory and able to perform light or sedentary work.
  2. Ambulatory and capable of all self-care; unable to work; up and about >50% of hours awake.
  3. Capable of limited self-care; confined to bed/chair >50% of hours awake.
  4. Completely disabled. Totally confined to bed or chair.
  5. Dead.
  Participants
    0-1 | 28 | 28 | 56
    2 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade ≥2 Radiation Dermatitis at 50 Gy (Per Protocol Set)
Description: Radiation dermatitis has been assessed according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4.03.
Time Frame: at 50 Gy (about 5 weeks)
Population: Per Protocol Set
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Treatment With Mepitel® Film: Patients treated with Mepitel® Film who were evaluable for radiation dermatitis at 50 Gy of radiotherapy and were treated per protocol.
- Arm B: Treatment With Standard Care: Patients treated with Standard Skin Care who were evaluable for radiation dermatitis at 50 Gy of radiotherapy and were treated per protocol.
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care
Number analyzed (Participants) | 9 | 27
Participants
  grade ≥2 radiation dermatitis | 3 | 9
  no grade ≥2 radiation dermatitis | 6 | 18

2. Secondary Outcome: Number of Participants With Grade ≥2 Radiation Dermatitis at 60 Gy (Per Protocol Set)
Description: as for outcome 1
Time Frame: at 60 Gy (about 6 weeks)
Population: Per Protocol Set
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Treatment With Mepitel® Film: Patients treated with Mepitel® Film who were evaluable for radiation dermatitis at 60 Gy of radiotherapy and were treated per protocol.
- Arm B: Treatment With Standard Care: Patients treated with Standard Skin Care who were evaluable for radiation dermatitis at 60 Gy of radiotherapy and were treated per protocol.
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care
Number analyzed (Participants) | 7 | 26
Participants
  grade ≥2 radiation dermatitis | 4 | 15
  no grade ≥2 radiation dermatitis | 3 | 11

3. Secondary Outcome: Number of Participants With Grade ≥3 Radiation Dermatitis at 50 Gy (Per Protocol Set)
Description: as for outcome 1
Time Frame: at 50 Gy (about 5 weeks)
Population: Per Protocol Set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care
Number analyzed (Participants) | 9 | 27
Participants
  grade ≥3 radiation dermatitis | 0 | 0
  no grade ≥3 radiation dermatitis | 9 | 27

4. Secondary Outcome: Number of Participants With Grade ≥3 Radiation Dermatitis at 60 Gy (Per Protocol Set)
Description: as for outcome 1
Time Frame: at 60 Gy (about 6 weeks)
Population: Patients of the Per Protocol Set who were evaluable for radiation dermatitis at 60 Gy.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care
Number analyzed (Participants) | 7 | 26
Participants
  grade ≥3 radiation dermatitis | 1 | 3
  no grade ≥3 radiation dermatitis | 6 | 23

5. Secondary Outcome: Number of Participants With Grade ≥2 Radiation Dermatitis at 50 Gy (Intention-to-treat Population)
Description: as for outcome 1
Time Frame: at 50 Gy (about 5 weeks)
Population: Intention-to-Treat Population
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Treatment With Mepitel® Film: Patients treated with Mepitel® Film who were evaluable for radiation dermatitis at 50 Gy of radiotherapy and belonged to the intention-to-treat population.
- Arm B: Treatment With Standard Care: Patients treated with Standard Skin Care who were evaluable for radiation dermatitis at 50 Gy of radiotherapy and belonged to the intention-to-treat population.
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care
Number analyzed (Participants) | 23 | 28
Participants
  grade ≥2 radiation dermatitis | 8 | 10
  no grade ≥2 radiation dermatitis | 15 | 18

6. Secondary Outcome: Number of Participants With Grade ≥2 Radiation Dermatitis at 60 Gy (Intention-to-treat Population)
Description: as for outcome 1
Time Frame: at 60 Gy (about 6 weeks)
Population: Patients of the Intention-To-Treat Population who were evaluable for radiation dermatitis at 60 Gy.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Treatment With Mepitel® Film: Patients treated with Mepitel® Film who were evaluable for radiation dermatitis at 60 Gy of radiotherapy and belonged to the intention-to-treat population.
- Arm B: Treatment With Standard Care: Patients treated with Standard Skin Care who were evaluable for radiation dermatitis at 60 Gy of radiotherapy and belonged to the intention-to-treat population.
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care
Number analyzed (Participants) | 23 | 27
Participants
  grade ≥2 radiation dermatitis | 15 | 16
  no grade ≥2 radiation dermatitis | 8 | 11

7. Secondary Outcome: Number of Participants With Grade ≥3 Radiation Dermatitis at 50 Gy (Intention-to-treat Population)
Description: as for outcome 1
Time Frame: at 50 Gy (about 5 weeks)
Population: Intention-To-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care
Number analyzed (Participants) | 23 | 28
Participants
  grade ≥3 radiation dermatitis | 0 | 0
  no grade ≥3 radiation dermatitis | 23 | 28

8. Secondary Outcome: Number of Participants With Grade ≥3 Radiation Dermatitis at 60 Gy (Intention-to-treat Population)
Description: as for outcome 1
Time Frame: at 60 Gy (about 6 weeks)
Population: Patients of the Intention-to-treat Population who were evaluable for radiation dermatitis at 60 Gy.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care
Number analyzed (Participants) | 23 | 27
Participants
  grade ≥3 radiation dermatitis | 1 | 3
  no grade ≥3 radiation dermatitis | 22 | 24

9. Secondary Outcome: Median Number of Radiation Fractions Until Occurence of Grade 2 Dermatitis
Description: The number of fractions of radiotherapy up to 50 Gy (50 Gy = 25 fractions) was counted in the intent-to-treat population, until grade 2 radiation dermatitis occurred.
Time Frame: up to 50 Gy (about 5 weeks)
Population: Patients of the Intention-to-treat Population who were evaluable for median number of radiation fractions (up to 50 Gy) until occurence of grade 2 dermatitis
Measure: Median (Full Range); unit: number of fractions of radiotherapy
Groups:
- Arm A: Treatment With Mepitel® Film: Patients treated with Mepitel® Film who were evaluable for radiation dermatitis up to 50 Gy of radiotherapy and belonged to the intention-to-treat population.
- Arm B: Treatment With Standard Care: Patients treated with Standard Skin Care who were evaluable for radiation dermatitis up to 50 Gy of radiotherapy and belonged to the intention-to-treat population.
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care
Number analyzed (Participants) | 23 | 28
number of fractions of radiotherapy | 23 [19 to 25] | 23 [9 to 25]

10. Secondary Outcome: Median Pain Score at the Irradiated Skin at 50 Gy
Description: The pain score will be assessed by using a numeric self rating scale from 0 (no pain) to 10 (maximum pain) points.
Time Frame: at 50 Gy (about 5 weeks)
Population: Patients of the Intention-to-treat Population who were evaluable for pain at 50 Gy.
Measure: Median (Full Range); unit: score on a scale
Groups:
- Arm A: Treatment With Mepitel® Film: Patients treated with Mepitel® Film who were evaluable for pain at baseline and at 50 Gy of radiotherapy and belonged to the intention-to-treat population.
- Arm B: Treatment With Standard Care: Patients treated with Standard Skin Care who were evaluable for pain at baseline and at 50 Gy of radiotherapy and belonged to the intention-to-treat population.
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care
Number analyzed (Participants) | 21 | 28
score on a scale | 0.0 [0 to 7] | 0.0 [0 to 7]

11. Secondary Outcome: Median Pain Score at the Irradiated Skin at 60 Gy
Description: The pain score will be assessed by using a numeric self rating scale from 0 (no pain) to 10 (maximum pain) points.
Time Frame: at 60 Gy (about 6 weeks)
Population: Patients of the Intention-to-treat Population who were evaluable for pain at 60 Gy.
Measure: Median (Full Range); unit: score on a scale
Groups:
- Arm A: Treatment With Mepitel® Film: Patients treated with Mepitel® Film who were evaluable for pain at baseline and at 60 Gy of radiotherapy and belonged to the intention-to-treat population.
- Arm B: Treatment With Standard Care: Patients treated with Standard Skin Care who were evaluable for pain at baseline and at 60 Gy of radiotherapy and belonged to the intention-to-treat population.
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care
Number analyzed (Participants) | 19 | 26
score on a scale | 2.0 [0 to 6] | 2.5 [0 to 8]

12. Secondary Outcome: Change in Quality of Life Between Screening and 50 Gy of Radiotherapy
Description: Quality of Life was assessed using the EORTC QLQ-C30 and QLQ-H&N35 questionnaires.
  For QLQ-C30, scoring of global health status and functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning) were assessed. Scores ranged from 0 to 100. A higher score represented a higher level of quality of life (global health status) and a higher level of functioning (functional scales).
  For QLQ-H&N35, symptom scales (pain, problems with swallowing, senses problems, speech problems, trouble with social eating, trouble with social contact) were assessed Scores ranged from 0 to 100. A higher score represented a higher level of symptomatology/problems.
  For both questionnaires (QLQ-C30 and QLQ-H&N35), the change between baseline and follow up at 50 Gy for each item was calculated by using the mean value of the differences between both time points of the evaluable patients.
Time Frame: at 50 Gy (about 5 weeks)
Population: For evaluations with the QLQ-C30 questionnaire, data of 19 patients (3 in Arm A, 16 in Arm B) were available, and for evaluations with the QLQ-H&N35 questionnaire, data of 18 patients (3 in Arm A, 15 in Arm B).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arm A: Treatment With Mepitel® Film: Patients treated with Mepitel® Film who were evaluable for quality of life at baseline and at 50 Gy of radiotherapy.
- Arm B: Treatment With Standard Care: Patients treated with Standard Skin Care who were evaluable for quality of life at baseline and at 50 Gy of radiotherapy.
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care
Number analyzed (Participants) | 3 | 16
score on a scale
  Change in global health status | 11.11 (12.73) | 19.79 (16.07)
  Change in physical functioning | -2.22 (7.70) | -15.0 (18.14)
  Change in role functioning | 0.0 (16.67) | -16.67 (23.57)
  Change in cognitive functioning | 0.0 (0.0) | -4.17 (20.64)
  Change in emotional functioning | -5.56 (9.62) | -3.65 (19.95)
  Change in social functioning | -16.67 (23.57) | 1.04 (26.15)
  Change regarding pain: number analyzed (Participants) | 3 | 15
  Change regarding pain | -19.44 (19.25) | -30.0 (30.67)
  Change regarding problems with swallowing: number analyzed (Participants) | 3 | 15
  Change regarding problems with swallowing | -13.89 (4.81) | -26.11 (34.20)
  Change regarding senses problems: number analyzed (Participants) | 3 | 15
  Change regarding senses problems | -22.22 (34.69) | -37.78 (33.61)
  Change regarding speech problems: number analyzed (Participants) | 3 | 15
  Change regarding speech problems | -7.41 (12.83) | -17.04 (13.36)
  Change regarding trouble with social eating: number analyzed (Participants) | 3 | 15
  Change regarding trouble with social eating | -5.56 (20.97) | -20.24 (23.98)
  Change regarding trouble with social contact: number analyzed (Participants) | 3 | 15
  Change regarding trouble with social contact | -2.22 (3.85) | -1.89 (8.79)

ADVERSE EVENTS:
Time Frame: up to 10 weeks following the start of radiotherapy
Arm/Group | Arm A: Treatment With Mepitel® Film | Arm B: Treatment With Standard Care
All-Cause Mortality (participants affected / at risk) | 2/28 | 1/29
Serious Adverse Events (participants affected / at risk) | 6/28 | 11/29
Other Adverse Events (participants affected / at risk) | 27/28 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Treatment With Mepitel® Film (N=28) | Arm B: Treatment With Standard Care (N=29)
Pheochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Severe dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Mucositis (Gastrointestinal disorders) | 1 | 1
Sepsis (Infections and infestations) | 1 | 2
Anemia (Blood and lymphatic system disorders) | 1 | 1
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 | 2
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Acute renal failure (Renal and urinary disorders) | 1 | 0
Methadon overdose (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
Creatinine increased (Renal and urinary disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Treatment With Mepitel® Film (N=28) | Arm B: Treatment With Standard Care (N=29)
Anemia (Blood and lymphatic system disorders) | 1 | 1
whte blood cell decreased (Investigations) | 1 | 1
impaired kidney function (Renal and urinary disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 1
Distress due to study product/procedure (Injury, poisoning and procedural complications) | 8 | 0
Feeling of tightness/suffcoating due to study product/procedure (Injury, poisoning and procedural complications) | 5 | 0
Radiation dermatitis (any grade) (Injury, poisoning and procedural complications) | 25 | 29
Radiation dermatitis (grade >=2) (Injury, poisoning and procedural complications) | 17 | 21
Mucositis (any grade) (Injury, poisoning and procedural complications) | 24 | 28
Mucositis (grade >=2) (Injury, poisoning and procedural complications) | 16 | 20
Taste disorders (any grade) (Injury, poisoning and procedural complications) | 16 | 24
Taste disorders (grade >=2) (Injury, poisoning and procedural complications) | 12 | 16
Xerostomia (any grade) (Injury, poisoning and procedural complications) | 17 | 26
Xerostomia (grade >=2) (Injury, poisoning and procedural complications) | 7 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT03047174/Prot_SAP_000.pdf